CLINICAL TRIAL: NCT00949325
Title: Phase I/II Trial of Torisel and Liposomal Doxorubicin in Patients With Advanced Soft Tissue and Bone Sarcomas
Brief Title: Safety and Efficacy Study of Torisel and Liposomal Doxorubicin for Patients With Recurrent Sarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Comprehensive Cancer Network (Network); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0963; NA_00028490 (Other: JHMI-IRB)
Record Dates: First submitted 2009-07-28; First posted 2009-07-30 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Sarcoma
Keywords: osteosarcoma; soft tissue sarcoma; rhabdomyosarcoma; leiomyosarcoma; Ewing's sarcoma; chondrosarcoma; liposarcoma; malignant fibrous histiocytoma; malignant peripheral nerve sheath tumor; pleiomorphic sarcoma; spindle cell sarcoma; synovial sarcoma; cancer stem cell
MeSH Terms: conditions — Sarcoma; Osteosarcoma; Rhabdomyosarcoma; Leiomyosarcoma; Sarcoma, Ewing; Chondrosarcoma; Liposarcoma; Histiocytoma, Malignant Fibrous; Neurofibrosarcoma; Sarcoma, Synovial | interventions — temsirolimus; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- temsirolimus plus liposomal doxorubicin (Experimental): Single arm study: Dose escalation of temsirolimus plus constant dose of liposomal doxorubicin.
  Interventions: Drug: temsirolimus plus liposomal doxorubicin

INTERVENTIONS:
Drug: temsirolimus plus liposomal doxorubicin — Patients were treated with temsirolimus (Torisel) weekly by IV and with liposomal doxorubicin (Doxil) (standard dose) by IV once every 28 days. Cohorts of patients receive sequentially increasing dose of temsirolimus until dose limiting toxicity (DLT) occurred and the maximally tolerated dose (MTD) was identified. The MTD dose was the standard dose of temsirolimus used for the remainder of the study. Dose modifications were based on protocol parameters for toxicities.
  Other Names: Torisel; Doxil

SUMMARY:
The purpose of this study is to identify a safe dosing regimen for the combination of Torisel and liposomal doxorubicin in patients with recurrent sarcoma. A secondary purpose of the study is to determine how effective this combination is for the treatment of recurrent sarcoma.

DETAILED DESCRIPTION:
The effectiveness of treatments for recurrent sarcomas is quite limited. One hypothesis to explain the refractory nature of recurrent sarcomas is the existence of chemotherapy-resistant sarcoma stem cells.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed sarcoma that is recurrent or refractory to conventional treatment
* Measurable disease by RECIST criteria
* ECOG (Eastern Cooperative Oncology Group) performance status < 2 (or Lansky/Karnofsky > 60% for children)
* Life expectancy greater than 3 months
* Adequate organ function
* absolute neutrophil count at least 1,500
* platelets at least 100,000
* bilirubin less than 1.5 x upper limit of normal
* AST (aspartate aminotransferase) and ALT(alanine aminotransferase) less than 2.5 x upper limit of normal
* creatinine less than 1.5 x upper limit of normal OR creatinine clearance at least 60 ml/min/1.73 m2
* fasting serum cholesterol less than 350
* fasting serum triglycerides less than 400
* PT (prothrombin) or INR (international normalized ratio) less than 1.3 x upper limit of normal
* normal urinalysis
* Ability to understand and sign the informed consent document

Exclusion Criteria:

* Prior chemotherapy or radiotherapy within 3 weeks of entering the study (6 weeks for nitrosoureas or mitomycin C)
* Prior treatment with a tyrosine kinase inhibitor within 10 days of entering the study
* History of pulmonary hypertension or pneumonitis
* Patients may not be receiving other investigational agents
* Prior therapy with rapamycin, rapamycin analogues, or tacrolimus
* Uncontrolled brain metastases
* History of grade 3 or 4 hypersensitivity to macrolide antibiotics
* Concurrent treatment with immunosuppressive agents other than a stable (for more than 2 weeks) dose of corticosteroids
* Uncontrolled intercurrent illness
* Pregnancy or breast feeding
* HIV-positive patients on combination antiretroviral therapy
* Grade 3 or 4 proteinuria

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Loeb, MD, PhD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Result] Thornton KA, Chen AR, Trucco MM, Shah P, Wilky BA, Gul N, Carrera-Haro MA, Ferreira MF, Shafique U, Powell JD, Meyer CF, Loeb DM. A dose-finding study of temsirolimus and liposomal doxorubicin for patients with recurrent and refractory bone and soft tissue sarcoma. Int J Cancer. 2013 Aug 15;133(4):997-1005. doi: 10.1002/ijc.28083. Epub 2013 Mar 4. PMID 23382028
- [Derived] Trucco MM, Meyer CF, Thornton KA, Shah P, Chen AR, Wilky BA, Carrera-Haro MA, Boyer LC, Ferreira MF, Shafique U, Powell JD, Loeb DM. A phase II study of temsirolimus and liposomal doxorubicin for patients with recurrent and refractory bone and soft tissue sarcomas. Clin Sarcoma Res. 2018 Nov 5;8:21. doi: 10.1186/s13569-018-0107-9. eCollection 2018. PMID 30410720

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1, Dose Level 3: Temsirolimus 15 mg/m^2
- Cohort 2, Dose Level 4: Temsirolimus 20 mg/m^2;
- Cohort 3, Dose Level 5: Temsirolimus 27mg/m^2
Period: Overall Study
Arm/Group | Cohort 1, Dose Level 3 | Cohort 2, Dose Level 4 | Cohort 3, Dose Level 5
Started | 3 | 18 | 3
Completed | 3 | 16 | 3
Not Completed | 0 | 2 | 0
Not completed — Adverse Event | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Temsirolimus Plus Liposomal Doxorubicin: Single arm consists of temsirolimus (Torisel) plus liposomal doxorubicin (Doxil). Temsirolimus is administered IV in sequentially escalating cohorts at doses between 15 and 50 mg/M2 (body surface area), once weekly. Liposomal doxorubicin is administered IV at 30 mg per M2 (body surface area) once every 28 days. Treatment may continue with both drugs for 2 years. Temsirolimus may continue beyond 2 years.
  temsirolimus plus liposomal doxorubicin: Patients will be treated with temsirolimus (Torisel) temsirolimus weekly by iv and with liposomal doxorubicin (Doxil) (standard dose) by iv once every 28 days. Cohorts of patients receive sequentially increasing dose of temsirolimus until maximally tolerated dose (MTD) is reached. Once MTD (standard dose) is achieved, dosing will be with standard doses for each drug, but dosing will be modified based on toxicity.
Arm/Group | Temsirolimus Plus Liposomal Doxorubicin
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 17
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 39.5 [9 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Incidence of Dose Limiting Toxicities
Description: Dose limiting toxicities in each dose cohort.
Time Frame: End of second 28-day cycle
Measure: Number; unit: participants
Groups:
- Number of Subjects Who Experienced Dose-Limiting Toxicities: Single arm consists of temsirolimus (Torisel) plus liposomal doxorubicin (Doxil). Temsirolimus is administered IV in sequentially escalating cohorts at doses between 15 and 50 mg/M2 (body surface area), once weekly. Liposomal doxorubicin is administered IV at 30 mg per M2 (body surface area) once every 28 days. Treatment may continue with both drugs for 2 years. Temsirolimus may continue beyond 2 years.
  temsirolimus plus liposomal doxorubicin: Patients will be treated with temsirolimus (Torisel) temsirolimus weekly by iv and with liposomal doxorubicin (Doxil) (standard dose) by iv once every 28 days. Cohorts of patients receive sequentially increasing dose of temsirolimus until maximally tolerated dose (MTD) is reached. Once MTD (standard dose) is achieved, dosing will be with standard doses for each drug, but dosing will be modified based on toxicity.
Arm/Group | Number of Subjects Who Experienced Dose-Limiting Toxicities
Number analyzed (Participants) | 24
participants
  Temsirolimus 15 mg/m^2 | 1
  Temsirolimus 20 mg/m^2 | 4
  Temsirolimus 27 mg/m^2 | 3

2. Primary Outcome: Part 2: Median Overall Survival of Subjects Who Were Treated at the Temsirolimus MTD, 20 mg/m^2
Description: Number of days from day 1 of treatment until date of death from any cause.
Time Frame: up to 5 years
Population: The number of analyzed participants does not include the 2 participants treated at the MTD who stopped treatment for early disease-related adverse events.
Measure: Median (Full Range); unit: days
Groups:
- Subjects Who Were Treated at the Temsirolimus MTD, 20 mg/m^2: Subjects who received Temsirolimus MTD, 20 mg/m^2 in Phase I of the study and all subjects in the Phase II study were included. from both Phase I and Phase II of the study are included.
Arm/Group | Subjects Who Were Treated at the Temsirolimus MTD, 20 mg/m^2
Number analyzed (Participants) | 16
days | 254 [50 to 1532]

3. Secondary Outcome: Median Progression-free Survival of Subjects Who Were Treated at the Temsirolimus MTD, 20 mg/m^2
Description: Interval from Date of start of treatment to date of disease progression or death from any cause. Disease progression is defined as at least 20% increase in sum of longest diameter of target lesions or appearance of any new lesions. Subjective determination of significant worsening of disease-related symptoms was considered clinical disease progression.
Time Frame: up to 3 years
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Groups:
- Subjects Who Were Treated at the Temsirolimus MTD, 20 mg/m^2: Subjects who received Temsirolimus MTD, 20 mg/m^2 in Phase I of the study and all subjects in the Phase II study were included from both Phase I and Phase II of the study who were not taken off study for early toxicity were included. Two of the eighteen subjects who were treated at the MTD were excluded.
Arm/Group | Subjects Who Were Treated at the Temsirolimus MTD, 20 mg/m^2
Number analyzed (Participants) | 16
days | 74 [7 to 797]

4. Secondary Outcome: Objective Response Rate
Description: Number of participants who completed at least 2 treatment cycles with evidence of response. Response is defined by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progression, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression
Time Frame: up to 5 years
Population: Only participants who completed at least 2 treatment cycles (14/18 participants) were included to assess this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Temsirolimus 20 mg/m^2 and 27 mg/m^2: Subjects who completed at least 2 cycles of treatment with temsirolimus dose of 20 mg/m^2 or 27 mg/m^2 were assessed for radiologic response.
Arm/Group | Temsirolimus 20 mg/m^2 and 27 mg/m^2
Number analyzed (Participants) | 14
Participants
  CR | 0
  PR | 1
  SD | 8
  PD | 5

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Whole blood temsirolimus and sirolimus levels were measured by LC/MS/MS
Time Frame: Prior to the initial dose on day 1, then 2, 6, and 24 hours post dose; prior to first dose of Cycle 2, then at 1, 2, 6, 24, 96, and 120 hours post dose in patients treated at the recommended phase 2 dose, Dose Level 4.
Population: Seven subjects had complete series of blood samples available for evaluation for both Temsirolimus, the parent drug and Sirolimus, the active metabolite. The number (N) evaluable participants is less than the number of participants from whom samples were collected due to inadvertent processing mishaps.
Measure: Mean (Standard Deviation); unit: mg/mL
Groups:
- Temsirolimus- Parent Drug: Whole blood temsirolimus and sirolimus levels were measured by LC/MS/MS
- Sirolimus- Active Metabolite: Whole blood temsirolimus and sirolimus levels were measured by LC/MS/MS. Cmax of Sirolimus was calculated using a non-compartmental model.
Arm/Group | Temsirolimus- Parent Drug | Sirolimus- Active Metabolite
Number analyzed (Participants) | 7 | 7
mg/mL | 346.2 (250) | 69.6 (23.2)

6. Secondary Outcome: Area Under the Curve (AUC)
Description: AUC was calculated using a single compartment model.
Time Frame: as for outcome 5
Population: Seven subjects had complete series of blood samples available for evaluation for both Temsirolimus, the parent drug and Sirolimus, the active metabolite. The analysis was per protocol. The number (N) evaluable samples is less than the number of collected samples due to inadvertent processing mishaps.
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Groups:
- Temsirolimus- Parent Drug: Whole blood temsirolimus and sirolimus levels were measured by LC/MS/MS. AUC was calculated using a single compartment model.
- Sirolimus- Active Metabolite: Whole blood temsirolimus and sirolimus levels were measured by LC/MS/MS. AUC was calculated using a single non- compartment model.
Arm/Group | Temsirolimus- Parent Drug | Sirolimus- Active Metabolite
Number analyzed (Participants) | 7 | 7
ng*hr/ml | 1210 (340) | 7499 (4591.1)

7. Secondary Outcome: Drug Clearance
Description: Whole blood temsirolimus and sirolimus levels were measured by LC/MS/MS.
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: L/hr/m2
Groups:
- Temsirolimus- Parent Drug: Clearance was calculated using a single compartment model.
Arm/Group | Temsirolimus- Parent Drug | Sirolimus- Active Metabolite
Number analyzed (Participants) | 7 | 7
L/hr/m2 | 17.8 (7.1) | NA (NA) — Values are not available. Drug clearance was not assessed in the Sirolimus-Active Metabolite arm.

8. Secondary Outcome: Mean Progression Free Survival of Subjects Who Were Treated at the Temsirolimus MTD, 20 mg/m^2
Description: Interval from start of treatment to disease progression or death from any cause. Disease progression is defined as at least 20% increase in sum of longest diameter of target lesions or appearance of any new lesions. Subjective determination of significant worsening of disease-related symptoms was considered clinical disease progression
Time Frame: up to 3 years
Measure: Mean (Full Range); unit: Days
Groups:
- Subjects Who Received Temsirolimus MTD, 20 mg/m^2: All subjects who received at least one dose of temsirolimus at the MTD, 20 mg/M^2 plus liposomal doxorubicin were included.
Arm/Group | Subjects Who Received Temsirolimus MTD, 20 mg/m^2
Number analyzed (Participants) | 16
Days | 195 [7 to 797]

9. Secondary Outcome: Mean Overall Survival of Subjects Who Were Treated at the Temsirolimus MTD, 20 mg/m^2
Time Frame: up to 5 years
Population: Subjects who received Temsirolimus MTD, 20 mg/m^2 in Phase I of the study and all subjects in the Phase II study were included from both Phase I and Phase II of the study are included.
Measure: Mean (Full Range); unit: Days
Groups:
- Subjects Who Were Treated at the Temsirolimus MTD, 20 mg/m^2: All subjects who received at least one dose of temsirolimus at the MTD, 20 mg/M^2 plus liposomal doxorubicin were included.
Arm/Group | Subjects Who Were Treated at the Temsirolimus MTD, 20 mg/m^2
Number analyzed (Participants) | 16
Days | 632 [50 to 1532]

10. Secondary Outcome: Time to Response
Description: Number of days after 2 cycles of treatment, until maximal response is observed.
Time Frame: up to 5 years
Population: Although the original protocol specified that "time to maximal response" would be an outcome measure that would be obtained, appropriate data were not collected, so this outcome measure cannot be evaluated or reported.
Arm/Group | Subjects Who Were Treated at the Temsirolimus MTD, 20 mg/m^2
Number analyzed (Participants) | 0

11. Secondary Outcome: Duration of Response
Description: Number of days until documentation of disease progression or date of death from other cause
Time Frame: up to 5 years
Population: Although the original protocol specified that "duration of response" would be an outcome measure that would be obtained, appropriate data were not collected, so this outcome measure cannot be evaluated or reported.
Arm/Group | Subjects Who Were Treated at the Temsirolimus MTD, 20 mg/m^2
Number analyzed (Participants) | 0

12. Secondary Outcome: Clinical Benefit Rate
Description: Number of days from documented improvement to disease progression.
Time Frame: up to 5 years
Population: Although the original protocol specified that "clinical benefit rate" would be an outcome measure that would be obtained, appropriate data were not collected, so this outcome measure cannot be evaluated or reported.
Arm/Group | Subjects Who Were Treated at the Temsirolimus MTD, 20 mg/m^2
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Temsirolimus Plus Liposomal Doxorubicin
Serious Adverse Events (participants affected / at risk) | 7/24
Other Adverse Events (participants affected / at risk) | 13/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temsirolimus Plus Liposomal Doxorubicin (N=24)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Required hospitalization.
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Required hospitalization.
Plural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Required hospitalization.
Respiratory failure (General disorders) | 2 (2) — death within 30 days of ending treatment x 2 subjects
Anorexia (Gastrointestinal disorders) | 1 (1) — Required hospitalization/feeding tube
Fever and chills (Infections and infestations) | 1 (1) — required hospitalization less than 30 days post treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temsirolimus Plus Liposomal Doxorubicin (N=24)
Neutropenia (Blood and lymphatic system disorders) | 5 (5)
anemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Elevated transaminases (Hepatobiliary disorders) | 2 (2)
Hyperlipedemia (Metabolism and nutrition disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Pancreatitis (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No